CLINICAL TRIAL: NCT02941237
Title: Development of a Robust and Reliable Pulse Oximeter for Use by Frontline Healthcare Providers Caring for Children With Pneumonia in Low-income Countries
Brief Title: Development of a Robust and Reliable Pulse Oximeter for Children With Pneumonia in Low-income Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Lifebox Foundation (Other)
Collaborators: Johns Hopkins University (Other); University College, London (Other); PACHI Malawi - Parent and Child Health Initiative Trust (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Isabeau Walker, Consultant Paediatric Anaesthetist, Honorary Senior Lecturer Great Ormond Street Hospital NHS Foundation Trust, The Lifebox Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPP1133291
Record Dates: First submitted 2016-10-16; First posted 2016-10-21 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Pneumonia in Children; Measurement of Peripheral Oxygen Saturation
Keywords: Pulse oximetry; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare worker measurement of SpO2 (Other): Measurement of SpO2 using the Lifebox pulse oximeter probe in children of different ages, stratified by age: 0-1 months, 2-11 months, 12-23 months and 24-59 months
  Interventions: Device: Pulse oximeter
- Expert measurement of SpO2 (Other): Measurement of SpO2 using the Lifebox pulse oximeter probe and Masimo oximeter probe in children of different ages, stratified by age: 0-1 months, 2-11 months, 12-23 months and 24-59 months
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — Time taken to measure oxygen saturation.
  Completion of usability questionnaire

SUMMARY:
This study is to test the usability of a new pulse oximeter probe designed for children 0-5 years.

DETAILED DESCRIPTION:
Pneumonia is the leading infectious cause of death in children under five. World Health Organization guidelines recommend measurement of peripheral oxygen saturation (SpO2) in children with pneumonia to guide treatment. This project focuses on the design of a new 'Lifebox' pulse oximeter probe for use in children 0-5 years of age.

A new oximeter probe compatible with the Lifebox oximeter has been designed to be used for children 0-5 years in all settings.

The aims of the study are to:

1. to evaluate the usability of the redesigned Lifebox oximeter probe by an expert user
2. to evaluate the usability of the redesigned oximeter probe by trained healthcare workers, against defined product specifications.
3. to compare the usability of the redesigned oximeter probe to a market leading probe

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

* Inpatients (or child awaiting surgery on pre-operative ward) in Great Ormond Street Hospital, or government facilities in Malawi and Bangladesh
* Aged 0 - 59 months
* Clinically stable (as judged by the ward sister and medical team)
* Parent (or adult with parental responsibility) present
* Informed consent from the parent (or adult with parental responsibility)

Healthcare worker participants:

* Nursing staff employed at Great Ormond Street Hospital who are trained in the use of pulse oximetry or government healthcare providers working in Malawi and Bangladesh
* Written informed consent from the healthcare worker

Exclusion Criteria:

Patient participants:

* Unstable or critically unwell patients (as judged by their medical team)
* Parents (or adult with parental responsibility) who are not able or willing to give informed consent
* Parents (or adult with parental responsibility) unable to speak English well enough to understand study methods or consent form (UK only)
* For part of the study assessing usability of the probe by healthcare workers, patients with oxygen saturation 95% or below will be excluded

Healthcare worker participants:

* Healthcare providers who are not trained to use a pulse oximeter
* Healthcare providers who have not given written informed consent

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 572 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Time to obtain SpO2 reading | Through completion of study, average one hour
  The time to obtain a stable reading will be declared by the healthcare worker or expert and noted by the independent observer, to give a proportion fulfilling the Target Product Profile (TPP).

OTHER OUTCOMES:
Usability questionnaire | Through study completion, average one hour
  Healthcare workers and the expert user will complete a usability questionnaire after completion of readings in children of different ages

CONTACTS AND LOCATIONS:
Overall Officials: Isabeau A Walker, FRCA, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (3):
- Sylhet hospital, Sylhet, Bangladesh
- District and referral hospitals, Lilongwe, Malawi
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burn SL, Chilton PJ, Gawande AA, Lilford RJ. Peri-operative pulse oximetry in low-income countries: a cost-effectiveness analysis. Bull World Health Organ. 2014 Dec 1;92(12):858-67. doi: 10.2471/BLT.14.137315. Epub 2014 Sep 24. PMID 25552770
- [Background] Finch LC, Kim RY, Ttendo S, Kiwanuka JK, Walker IA, Wilson IH, Weiser TG, Berry WR, Gawande AA. Evaluation of a large-scale donation of Lifebox pulse oximeters to non-physician anaesthetists in Uganda. Anaesthesia. 2014 May;69(5):445-51. doi: 10.1111/anae.12632. PMID 24738801
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Duke T, Wandi F, Jonathan M, Matai S, Kaupa M, Saavu M, Subhi R, Peel D. Improved oxygen systems for childhood pneumonia: a multihospital effectiveness study in Papua New Guinea. Lancet. 2008 Oct 11;372(9646):1328-33. doi: 10.1016/S0140-6736(08)61164-2. Epub 2008 Aug 15. PMID 18708248
- [Background] Bhutta ZA, Das JK, Walker N, Rizvi A, Campbell H, Rudan I, Black RE; Lancet Diarrhoea and Pneumonia Interventions Study Group. Interventions to address deaths from childhood pneumonia and diarrhoea equitably: what works and at what cost? Lancet. 2013 Apr 20;381(9875):1417-1429. doi: 10.1016/S0140-6736(13)60648-0. Epub 2013 Apr 12. PMID 23582723
- [Background] Matai S, Peel D, Wandi F, Jonathan M, Subhi R, Duke T. Implementing an oxygen programme in hospitals in Papua New Guinea. Ann Trop Paediatr. 2008 Mar;28(1):71-8. doi: 10.1179/146532808X270716. PMID 18318953
- [Background] Soofi S, Ahmed S, Fox MP, MacLeod WB, Thea DM, Qazi SA, Bhutta ZA. Effectiveness of community case management of severe pneumonia with oral amoxicillin in children aged 2-59 months in Matiari district, rural Pakistan: a cluster-randomised controlled trial. Lancet. 2012 Feb 25;379(9817):729-37. doi: 10.1016/S0140-6736(11)61714-5. Epub 2012 Jan 27. PMID 22285055
- [Background] Yeboah-Antwi K, Pilingana P, Macleod WB, Semrau K, Siazeele K, Kalesha P, Hamainza B, Seidenberg P, Mazimba A, Sabin L, Kamholz K, Thea DM, Hamer DH. Community case management of fever due to malaria and pneumonia in children under five in Zambia: a cluster randomized controlled trial. PLoS Med. 2010 Sep 21;7(9):e1000340. doi: 10.1371/journal.pmed.1000340. PMID 20877714
- [Background] Faulkner L. Beyond the five-user assumption: benefits of increased sample sizes in usability testing. Behav Res Methods Instrum Comput. 2003 Aug;35(3):379-83. doi: 10.3758/bf03195514. PMID 14587545
- [Derived] King C, Boyd N, Walker I, Zadutsa B, Baqui AH, Ahmed S, Islam M, Kainja E, Nambiar B, Wilson I, McCollum ED. Opportunities and barriers in paediatric pulse oximetry for pneumonia in low-resource clinical settings: a qualitative evaluation from Malawi and Bangladesh. BMJ Open. 2018 Jan 30;8(1):e019177. doi: 10.1136/bmjopen-2017-019177. PMID 29382679
- See also: Description of usability testing from the British Standards Institute — http://www.bsigroup.com/LocalFiles/EN-AU/ISO%2013485%20Medical%20Devices/Whitepapers/The%20growing%20role%20of%20human%20factors%20and%20usability%20engineering%20for%20medical%20devices.pdf
- See also: Guidance from British Standards Institute on best practices in usability testing — http://www.bsigroup.com/meddev/LocalFiles/en-US/Roadshow%20Resources%202015/Fall/Usability%20best%20practices.pdf

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT02941237/Prot_SAP_000.pdf
  • Informed Consent Form: Parent Consent (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT02941237/ICF_001.pdf
  • Informed Consent Form: HealthCare Worker Consent (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT02941237/ICF_002.pdf